CLINICAL TRIAL: NCT05553860
Title: Two Cohort Prospective Single Blinded Patient Crossover Trial Comparing Anterior Protrusive and Sibilant Phoneme Mandibular Positioning Techniques for Dental Sleep Appliances
Brief Title: Comparing Two Mandibular Positioning Techniques for Dental Sleep Appliances
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00097563
Record Dates: First submitted 2022-09-21; First posted 2022-09-23 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Sleep Apnea, Obstructive; Occlusal Splints
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anterior Protrusive (Active Comparator): use of anterior protrusive positioning technique
  Interventions: Other: Speech positioning technique
- Speech Position (Experimental): use of speech positioning technique
  Interventions: Other: Speech positioning technique

INTERVENTIONS:
Other: Speech positioning technique — Speech positioning technique

SUMMARY:
This is a prospective study that directly compares the use of speech vs an anterior protrusive technique for mandibular positioning.

DETAILED DESCRIPTION:
Obstructive sleep apnea is a medical condition where a person has great difficulty with breathing, or stops breathing all together, while asleep. This is a medical condition for which one of the current standard treatments is the use of a custom-made dental appliance to help hold the person's airway open while asleep so that the person does not suffocate while sleeping. Current methodology within dentistry is to position the mandible based on the person's maximum ability to position their mandible forward as the starting point and then slowly move the bottom jaw forward as necessary. Recent literature has shown that different mandibular positioning techniques may require less protrusion, less titrations, and potentially decreased side effects compared with the traditional protrusive techniques. One of the most promising techniques involves the use of speech to determine mandibular position. This technique would not require that a patient place their jaw outside of their normal functional range and could potentially decrease the face pain/jaw joint problems commonly associated with the use of oral sleep appliances for the treatment of obstructive sleep apnea. The use of speech as the determinant for where to position the mandible is important for muscular balance. Minimal research has been done in this area, with most studies being either retrospective or confounded by other variables. This will be the first prospective study that directly compares the use of speech vs an anterior protrusive technique for mandibular positioning.

ELIGIBILITY:
Inclusion Criteria:

Patient diagnosed with obstructive sleep apnea, and

* Prescription/order for a dental sleep appliance
* 18 years or older
* Treatment planned in accordance with AADSM treatment guidelines

Exclusion Criteria:

* There are no separate exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-12-05 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Apnea-hypopnea index (AHI) | 3 months
  Measurement to determine whether both mandibular positioning techniques provide similar management of obstructive sleep apnea

SECONDARY OUTCOMES:
Overjet | 3 months
  Measurement to determine whether there is a significant difference in final treatment mandibular position between the positioning techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Enoch Ng, DDS, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No